CLINICAL TRIAL: NCT04406220
Title: The Effect of Large Versus Small Clog Size on Healthcare Professional Emergency Response Time: a Randomized Controlled Trial
Brief Title: The Effect of Large Versus Small Clog Size on Emergency Response Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.J.S. de Grooth, MD, Coordinating investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-clog
Record Dates: First submitted 2020-03-02; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Clothing; Occupational Injuries
MeSH Terms: conditions — Occupational Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small clog size (Active Comparator)
  Interventions: Other: Small clog size
- Large clog size (Active Comparator)
  Interventions: Other: Large clog size

INTERVENTIONS:
Other: Small clog size — Participants will be randomized to run in small clogs
  Arms: Small clog size
Other: Large clog size — Participants will be randomized to run in large clogs
  Arms: Large clog size

SUMMARY:
In many hospitals, clogs, usually white, are provided for healthcare workers. In our hospital, health care professionals from the department of intensive care medicine may be summoned to an emergency situation on a 24/7 basis. Clogs are thought to be of importance for running. Although clogs are available in several sizes, clog size is typically left to the discretion of the individual healthcare worker. Interestingly,

The primary goal of this randomized controlled trial is to assess if wearing large size clogs as compared to small size clogs results in increased running speed.

Participants will be randomized to small versus large clog size using a using randomly permuted blocks stratified by gender. Following randomization, participants will wear the clogs of allocated size and complete a standardized running course.

The primary endpoint is the time taken to complete the course.

The enrolment of 50 subjects would provide 80% power to show a 5-second difference in the response time at an average response time of 30 seconds with a 6 second standard deviation.

The ethical committee judged the study protocol exempt from extensive review.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers aged 18 years or older.

Exclusion Criteria:

* Inability to run on clogs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Time to complete the running course | Follow-up until 60 minutes.
  The time to complete the course will be compared between the two groups using a linear model with the randomized allocation and the stratification variable as covariates.

SECONDARY OUTCOMES:
Adverse events | Follow-up until 60 minutes.
Time to complete the running course for specific subgroups: By gender, job function, level of fitness. | Follow-up until 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Elbers, MD, PhD, Study Chair — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elbers PWG, de Grooth HJ, Girbes ARJ. The effect of small versus large clog size on emergency response time: A randomized controlled trial. J Crit Care. 2020 Dec;60:116-119. doi: 10.1016/j.jcrc.2020.07.028. Epub 2020 Aug 8. PMID 32799180